CLINICAL TRIAL: NCT03299712
Title: Protocol for the Post-approval Study of Artefill for Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suneva Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 521-01; NCT00778531 (obsolete NCT alias)
Record Dates: First submitted 2014-11-17; First posted 2017-10-03 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Granulomatous Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArteFill (Other): This post-approval study will evaluate the continuing safety of ArteFill® as an injectable implant for correction of nasolabial folds over the course of five years post implantation, with a focus on determining the incidence of granuloma formation. Incidence of adverse events and subject satisfaction with respect to the subject's personal expectations will be assessed.
  Interventions: Device: ArteFill

INTERVENTIONS:
Device: ArteFill — soft tissue filler

SUMMARY:
This study is a five-year, multi-center, non-randomized, non-controlled post-approval study designed to follow a total of 1000 consecutive qualified and consenting subjects treated with ArteFill® in the course of clinical practice at approximately twenty-five centers and all subjects must have a previously documented negative skin test prior to receiving treatment. The incidence of granuloma formation will be monitored.

DETAILED DESCRIPTION:
This study is a multi-center, non-randomized, non-controlled post-approval study designed to follow a total of 1000 consecutive qualified and consenting subjects treated with ArteFill® in the course of clinical practice at approximately twenty-five centers. All potential qualifying subjects at a given site should be given the opportunity to participate in the study. Inclusion and exclusion criteria will be limited to those in the approved labeling for ArteFill® and treatment will be according to the approved product labeling. Subjects must have a previously documented negative skin test prior to treatment. Follow-up for subject-reported potential adverse events and satisfaction data will be by mail or telephone questionnaire survey every six months for the first two years after the final treatment session and then every year for a total of five years of follow-up. The subject will be contacted by his or her investigator if a problem is identified in the questionnaire response as reviewed by the Sponsor or their designee. Potential adverse events reported in the follow-up questionnaires will be investigated further by means of office visits, as necessary, or via telephone.

Adverse events will be confirmed and reported by the investigators. If an adverse event is determined by the investigator to possibly be a granuloma, it will be investigated via histology. If a subject for whom an adverse event is reported has received additional aesthetic or non-aesthetic treatment to the affected area, available information on such treatment will be collected and the subject will be continued to be followed per protocol. Such subjects will not be excluded from the analysis, but will be evaluated separately. Effectiveness data will be collected during the study and will consist of the subject's assessment of satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female 18 years of age or older.
2. Subject has provided written and verbal informed consent.
3. Subject is willing to comply with study instructions and return to the clinic for required visits.
4. Subject is willing to withhold additional aesthetic implant therapies to the NLF [e.g., other soft tissue fillers: Restylane, Silicone, Radiesse, Sculptra) or implants: gortex, silastic, thread lift, etc.] for the duration of the study.
5. Subject has a documented negative skin test.

Exclusion Criteria:

1. Subject has any skin pathology or condition that could interfere with the evaluation of the treatment areas.
2. Subject has a history of systemic granulomatous diseases active or inactive (e.g.

   Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (.e.g., lupus, dermatomyositis, etc.).
3. Subject is immuno-compromised in the opinion of the investigator because of disease or medical therapy (e.g., HIV, use of chemotherapy, etc.)
4. Subject has been treated with any of the following in their NLF in the time intervals specified prior to the start of their participation in the study:

   * Bovine collagen - 6 months
   * Porcine or human collagen - one year
   * Hyaluronic acid - one year
   * Hydroxylapatite - one year
   * Autologous fat - at any time
   * Polymethylmethacrylate or other acrylates - at any time
   * Polyacrylamide - at any time
   * Polyethylene oxide - at any time
   * Polylactic acid - at any time
   * Liquid silicone - at any time
   * Other permanent implant material (FDA approved or not) - at any time
5. Subject has had the placement of any surgical implants in the NL folds region (e.g., Gortex, Silastic implants, thread lifts, etc.) at any time.
6. Subject has a history of multiple severe allergies or allergies manifested by anaphylaxis.
7. Subject has a history of allergy to lidocaine.
8. Subject has a history of allergies to any bovine collagen products, including but not limited to injectable collagen, collagen implants, hemostatic sponges, and collagen-based sutures.
9. The subject has known hypersensitivity or previous allergic reaction to any of the components of the study devices not previously mentioned.
10. Subject is undergoing or planning to undergo desensitization injections to meat products.
11. Subject has any condition which, in the Investigator's opinion, would make it unsafe for the subject to participate in this research study.
12. Subject is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function.
13. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2007-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The incidence of granuloma formation. | 5 years
  To determine the incidence of granuloma formation.
Incidence of unanticipated adverse events | 5 years
  Safety will be assessed based on the incidence of serious unanticipated adverse events. Unanticipated adverse events will be characterized by the severity and relation to the implant product.
Incidence of anticipated adverse events | 5 years
  The incidence of anticipated adverse events will be assessed at each follow-up visit.

SECONDARY OUTCOMES:
Assess of subject satisfaction | 5 years
  Subjects assessed their satisfaction using the 5-point Likert Scale Subject Satisfaction Assessment Scale. This scale has the following measurements: 1- Very Satisfied, 2=Satisfied, 3=Somewhat Satisfied, 4= Dissatisfied and 5=Very Dissatisfied.